CLINICAL TRIAL: NCT02981290
Title: A Randomized, Open Label, Four-way Crossover Study to Compare the Pharmacokinetics of Mycophenolate Mofetil Metabolites From Four Tablet Formulations in Healthy Subjects
Brief Title: Study to Compare the Pharmacokinetics of Mycophenolate Mofetil Metabolites From Four Tablet Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WP21980
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Renodapt Then Mycept Then Cellmune Then CellCept (Experimental): Participants will receive Renodapt in first treatment period (each treatment period= 3 days) followed by Mycept in second treatment period then Cellmune in third treatment period and CellCept in fourth treatment period. A washout period of 7 days will be separating each treatment period.
  Interventions: Drug: Renodapt; Drug: Mycept; Drug: Cellmune; Drug: CellCept
- Mycept Then CellCept Then Renodapt Then Cellmune (Experimental): Participants will receive Mycept in first treatment period (each treatment period= 3 days) followed by CellCept in second treatment period then Renodapt in third treatment period and Cellmune in fourth treatment period. A washout period of 7 days will be separating each treatment period.
  Interventions: Drug: Renodapt; Drug: Mycept; Drug: Cellmune; Drug: CellCept
- Cellmune Then Renodapt Then CellCept Then Mycept (Experimental): Participants will receive Cellmune in first treatment period (each treatment period= 3 days) followed by Renodapt in second treatment period then CellCept in third treatment period and Mycept in fourth treatment period. A washout period of 7 days will be separating each treatment period.
  Interventions: Drug: Renodapt; Drug: Mycept; Drug: Cellmune; Drug: CellCept
- CellCept Then Cellmune Then Mycept Then Renodapt (Experimental): Participants will receive CellCept in first treatment period (each treatment period= 3 days) followed by Cellmune in second treatment period then Mycept in third treatment period and Renodapt in fourth treatment period. A washout period of 7 days will be separating each treatment period.
  Interventions: Drug: Renodapt; Drug: Mycept; Drug: Cellmune; Drug: CellCept

INTERVENTIONS:
Drug: Renodapt — Renodapt will be administered as 500 milligrams (mg) tablet orally on Day 1 in any treatment periods.
Drug: Mycept — Mycept will be administered as 500 mg tablet orally on Day 1 in any treatment periods.
Drug: Cellmune — Cellmune will be administered as 500 mg tablet orally on Day 1 in any treatment periods.
Drug: CellCept — CellCept will be administered as 500 mg tablet orally on Day 1 in any treatment periods.

SUMMARY:
This is a single center, randomized, open label, 4-treatment, 4-period, 4-sequence, 4-way crossover study to compare the pharmacokinetics of mycophenolate mofetil (MMF) metabolites from 4 tablet formulations in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

A body mass index (BMI) between 18 and 32 kilogram per meter square (kg/m^2)

Exclusion Criteria:

* Any evidence of clinically significant allergic, renal, cardiac, bronchopulmonary, vascular, gastro-intestinal, neurological, metabolic or immunodeficiency disorders, cancer, hepatitis or cirrhosis
* Any evidence of gall bladder surgery, surgery of the gastro-intestinal tract or any other medical condition considered likely to affect drug absorption
* Any major illness within 2 months prior to first dosing or febrile illness within 14 days prior to first dosing
* Any known history of clinically significant allergic reactions or drug hypersensitivity, especially hypersensitivity to MMF or mycophenolic acid (MPA)
* Any other ongoing concomitant disease or condition that could interfere with, or the treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participants
* Any prescribed or over-the-counter (OTC) medication, herbal medicine or dietary aid taken within 2 weeks before the first study drug dosing or within six times the elimination half-life of the medication before the first study drug dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)] of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Maximum Observed Plasma Concentration (Cmax) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Time to Reach Maximum Observed Plasma Concentration (Tmax) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Absorption Lag Time (Tlag) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Plasma Terminal Half-Life (t1/2) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Apparent Oral Clearance (CL/F) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1

SECONDARY OUTCOMES:
Apparent Oral Volume of Distribution (V/F) of MPA | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
AUC (0-inf) of the Glucuronide Metabolite of MPA (MPAG) | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
AUClast of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Cmax of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Tmax of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Tlag of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
t1/2 of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
CL/F of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
V/F of MPAG | Predose (0.5 hours), and 0.33, 0.66, 1, 1.33, 1.66, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose on Day 1
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch Clinical Studies Trust, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reigner B, Grange S, Bentley D, Banken L, Abt M, Hughes R, Scheubel E, Guentert TW. Generics in transplantation medicine: Randomized comparison of innovator and substitution products containing mycophenolate mofetil . Int J Clin Pharmacol Ther. 2019 Oct;57(10):506-519. doi: 10.5414/CP203487. PMID 31397274